CLINICAL TRIAL: NCT00160771
Title: University of Florida Biomechanics/Motion Analysis Laboratory Data Bank
Brief Title: Biomechanics/Motion Analysis Laboratory Data Bank
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201501196
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Kinematics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Joint Motion Analysis: Joint motion will be recorded for analysis.
  Interventions: Behavioral: Joint Motion Analysis

INTERVENTIONS:
Behavioral: Joint Motion Analysis — Joint motion will be recorded for analysis.
  Other Names: No other names

SUMMARY:
The purpose of the data bank is to collect data on joint motion.

DETAILED DESCRIPTION:
Biomechanical aspects, including ground reaction forces, range of motion of involved extremities, EMG data and videotape records of human motion will be collected and stored as part of the normal clinical care of patients seen in the UF Biomechanics/Motion Analysis Laboratory. All persons seen in motion analysis laboratory will be told of study and asked to participate. Those agreeing to participation will give informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Any person having joint analysis done for medical or personal need

Exclusion Criteria:

* None, any person having joint analysis done for medical or personal need and interested in participation will be asked to sign informed consent.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Biomechanical/Motion Analysis Laboratory
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2005-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Range of Motion values | one day
  Joint range of motion is measured in degrees for the hips, knees, ankles, shoulders and elbows

CONTACTS AND LOCATIONS:
Overall Officials: MaryBeth Horodyski, Ed.D., Principal Investigator — University of Florida
Locations (1):
- UF Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States